CLINICAL TRIAL: NCT04283721
Title: Optimal Method and Timing to Provide Information on Epidural and Spinal Anaesthesia for Primiparas: A Qualitative Randomised Control Trial
Brief Title: Optimal Method and Timing to Provide Information on Epidural and Spinal Anaesthesia for Primiparas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sligo General Hospital (Other)
Responsible Party: Principal Investigator, Omar Tujjar, Principal Investigator, Sligo General Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 786
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Patient Satisfaction; Confidence, Self
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No Video (No Intervention): These patients will not see the educational video on epidural/spinal analgesia and will receive the usual Irish standard of care.
- Antenatal Video (Experimental): These patients will see the educational video on epidural/spinal analgesia only at the antenatal classes.
  Interventions: Other: Educational video
- Labour Video (Experimental): These patients will see the educational video on epidural/spinal analgesia only at the beginning of labour.
  Interventions: Other: Educational video
- Video Twice (Experimental): These patients will see the educational video on epidural/spinal analgesia twice (during antenatal classes and at the beginning of labour).
  Interventions: Other: Educational video

INTERVENTIONS:
Other: Educational video — Ten-minutes educational video on epidural/spinal analgesia benefits and side effects (sample video link: https://youtu.be/jAhoKhvcbP4). The informational video will be administered by co-investigators, who are anaesthesiologists. The video will be shown on an institutional iPad that will be thoroughly disinfected by the co-investigators before and after each use. Co-investigators will receive training on the disinfection process, and each disinfection will be documented on a logbook, dated and signed by the co-investigators.
  Arms: Antenatal Video; Labour Video; Video Twice

SUMMARY:
Expectant mothers can give birth to their child either by vaginal delivery or by a caesarean section (the latter can be planned or necessary during an emergency). Among the pain-relieving options for vaginal delivery, they can choose to receive epidural analgesia. In case of a caesarean section, the three anaesthetic options are epidural, spinal, or general anaesthesia.

The current Irish standard of care for the provision of information and consent for epidural and spinal anaesthesia entails a consultation with the anaesthesiologists at the request of the expectant mothers, shortly before the procedure. The uniformity of the information provided with this method is being debated. Moreover, there is a lack of consensus on the best timing and setting to informing patients.

With the aim of standardising the provision of information on epidural and spinal anaesthesia, the Anaesthetic Department in Sligo University Hospital has created an informational video on such procedures, in which all benefits and possible complications are explained in detail.

This video can be shown to expectant mothers at the antenatal classes or in the early stage of labour, as soon as they present to the labour ward.

Importantly, this video is not aimed at promoting the use of the epidural catheter, rather at providing expectant mothers all the information on the technique, benefits, side effects and possible complications of the procedure.

The main objective of this study is to evaluate whether this informational video is effective in improving patient confidence and satisfaction regarding these pain-relieving options, and what is the optimal timing to show the video. Our hypothesis is that, compared to the control group, women who watch the informational video will feel more confident in choosing to receive or not these pain-relieving options and therefore have a more positive childbirth experience.

This study is a randomised control trial. Randomisation will produce 4 groups in total. Depending on the group allocation, participants may or may not be shown the informational video in relation to spinal/epidural anaesthesia at various stages (antenatal classes or at the time of their arrival on the labour ward). The control group will receive the usual Irish standard of care.

After delivery, the patients will be interviewed with a questionnaire that will explore:

* Their satisfaction with the information provided in relation to the epidural/spinal anaesthesia;
* Their confidence in choosing to receive/not to receive these pain relieving options;
* Their ability to recollect the information provided on these pain-relieving options.

To the extent of our knowledge, this is the first study that aims at improving parturients' sense of confidence and satisfaction in relation to the information provided on epidural and spinal anaesthesia. Should patients find this means of information beneficial to their care and overall experience, there is potential for nationwide distribution.

ELIGIBILITY:
Inclusion Criteria:

* Primiparas attending the labour ward in the early stage of labour

Exclusion Criteria:

* Patient refusal to participate
* Advanced phase of labour (as clinically assessed by midwives)
* Patient distress (as clinically assessed by midwives and anaesthesiologists)
* Intrauterine death
* Patients under 18 years of age
* Patients unable to provide consent
* Non-English speakers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2020-03-02 (Estimated); Primary Completion 2021-06-28 (Estimated); Study Completion 2021-06-28 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction through survey questionnaire. | 48 hours after delivery
  Women's satisfaction with the information received in relation to the epidural/spinal anaesthesia will be evaluated with a questionnaire developed with the help of a Consultant Psychiatrist. This questionnaire will be administered 48 hours after delivery.

SECONDARY OUTCOMES:
Patient confidence through survey questionnaire. | 48 hours after delivery
  Women's degree of confidence in choosing to receive or not to receive epidural/spinal as pain-relieving options will be evaluated with a questionnaire developed with the help of a Consultant Psychiatrist. This questionnaire will be administered 48 hours after delivery.
Patient recollection through survey questionnaire. | 48 hours after delivery
  Women's degree of recollecting the information received on epidural/spinal anaesthesia will be evaluated with a questionnaire developed with the help of a Consultant Psychiatrist. This questionnaire will be administered 48 hours after delivery.

IPD SHARING:
Plan to Share IPD: No